CLINICAL TRIAL: NCT02758756
Title: Pilot Study on Energy Therapy or Massage to Reduce Fatigue in Breast and Prostate Cancer Patients on Hormone Therapy
Brief Title: Pilot Study on Energy Therapy or Massage to Reduce Fatigue
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Rochester (Other)
Responsible Party: Principal Investigator, Luke Peppone, Assistant Professor, University of Rochester
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: UCCS15115
Record Dates: First submitted 2016-04-28; First posted 2016-05-02 (Estimated); Last update posted 2019-07-05 (Actual); Status verified 2019-07

CONDITIONS: Fatigue
MeSH Terms: conditions — Fatigue | interventions — Massage; Therapeutic Touch

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Massage (Active Comparator): Subjects assigned to Arm 1 will receive two massage treatments approximately two weeks apart.
  Interventions: Other: Massage
- Two Reiki Tx (Experimental): Subjects assigned to Arm 2 will receive two Reiki treatments approximately two weeks apart.
  Interventions: Other: Reiki
- Four Reiki Tx (Experimental): Subjects assigned to Arm 3 will receive four Reiki treatments approximately 1 week apart.
  Interventions: Other: Reiki

INTERVENTIONS:
Other: Massage — Treatments will be on a massage table and last up to 75 minutes. We do not specify what will occur during the massage treatments. Instead we will follow the model of relying on the professional expertise of the therapist in combination with input from the client to determine what should happen in the session. We specify that energy healing techniques not be used, because that is our research comparison condition. We also specify that conversation between the massage therapist and the patient be kept to the minimum necessary to effectively provide the treatment. This is not meant to be talk therapy.
  Arms: Massage
Other: Reiki — Reiki treatments will be provided by Reiki Masters on a massage table and last up to 75 minutes. We will not specify what will occur during the Reiki treatments. Instead we will follow the model of relying on the professional expertise of the therapist in combination with input from the client to determine what should happen in the session. That being said, we will ask that two specific things be kept to a minimum. The first is that we ask that Swedish massage techniques not be used, because that is our research comparison condition. The second is that conversation between the massage therapist and the patient be kept to the minimum necessary to effectively provide the treatment. This is not meant to be talk therapy.
  Other Names: Energy Therapy
  Arms: Four Reiki Tx; Two Reiki Tx

SUMMARY:
The proposed study will assess whether either massage or an Integrative Medicine practice called Reiki can alleviate fatigue in subjects receiving hormonal treatments. Reiki is classified by the National Center for Complementary and Integrative Health as a biofield/touch therapy, and Reiki practitioners believe that their gentle therapy promotes healing and well-being by unblocking and balancing energy flow and re-establishing homeostasis within the human energy field. The study is a three-arm randomized clinical trial in 99 breast and prostate cancer patients who are undergoing hormonal therapy (i.e., androgen deprivation therapy (ADT) for males or an aromatase inhibitor (AI) for females) and currently experiencing fatigue. Subjects will be studied during ten weeks of hormonal therapy with two weeks of baseline assessments followed by a four-week intervention, and a four-week post-intervention period. Arm 1: Subjects will receive two Swedish-style massages. Arm 2: Lower-dose Reiki intervention - Subjects will receive two Reiki treatments. Arm 3: Higher-dose Reiki intervention - Subjects will receive four Reiki treatments.

DETAILED DESCRIPTION:
5.1 This will be a randomized three-arm clinical trial pilot study of an intervention examining the efficacy of either massage or Reiki in reducing fatigue associated with hormonal treatment and to determine if four Reiki treatments are more effective than two in controlling fatigue. Subjects will be studied during ten weeks of hormonal therapy with two weeks of baseline assessments followed by a four-week intervention, and a four-week post-intervention period.

5.1.1 All ancillary treatments for control of symptoms caused by the cancer or its treatment may be administered as clinically indicated.

5.1.2 The current protocol is for a pilot study designed to gather preliminary efficacy and feasibility data for the development of a planned RO1 submission. Our intention is to gather preliminary data to generate effect size estimates for power calculations for an anticipated RO1 application. We will also use this preliminary data to help us determine whether or not we should drop or modify one or more of the current study arms when designing the planned RO1 study.

5.1.3 It is preferred that the study be completed in a time-span of ten calendar weeks, however if the subject or practitioner is unable to attend an appointment during a scheduled week, that week will not count as a study week, and it will be designated a skipped week. Only two skipped weeks will be allowed, so the maximum length of the study will be twelve calendar weeks. Subjects will not complete questionnaires during skipped weeks, and skipped weeks may not be consecutive.

5.2 Consent Process and Assessment

5.2.1 After providing written informed consent (and receiving a signed copy), the subject will complete an On-Study Data Form providing demographic and clinical data. Questions concerning the subject's experience with both Reiki and massage (and related treatments) and expectations for their efficacy in relieving fatigue are also included. Subjects will also complete a quality of life (QOL) questionnaire and sleep quality (SQ) questionnaire at time of consent.

5.2.2 Subjects will be asked to completed study questionnaires at home. They will have the option of completing questionnaires via the REDCap online survey system (see Section 6.10) or on paper. If they choose to complete paper questionnaires, they will be given a packet of study questionnaires at the time of consent. The questionnaire packet will consist of seven sets of questionnaires. Each set will have the Brief Fatigue Inventory (BFI), the Insomnia Severity Index (ISI), and a Symptom Inventory. In addition, the sixth and seventh sets of questionnaires will also include the Pittsburgh Sleep Quality Inventory (PSQI) to assess SQ, the Functional Assessment of Chronic Illness Therapy-Fatigue (FACIT-F) to assess QOL, and the Profile of Mood States (POMS). If they choose to complete questionnaires via REDCap, they will be asked to complete the same questionnaires through the online survey system. Subjects electing to use REDCap will also be given one set of paper questionnaires to be used in the event that computer access is not available when needed.

5.2.3 Subjects will be asked to complete one set of questionnaires (either through REDCap or on paper) each Friday night of the 2-week baseline and the 4-week intervention period. They will be asked to complete a final set on Friday of Week 10. A set of questionnaires takes about 10-20 minutes to complete.

5.2.4 Reminder phone calls or emails will be made by study personnel each Friday to assist the subject in remembering to complete the study forms. If they have chosen to complete paper questionnaires, they will also be instructed to return them in the provided stamped, pre-addressed envelope. (Permission will be obtained to leave messages on a subject's voicemail before any messages are left.)

5.3 An optional Heart Rate Variability (HRV) assessment will be done during study weeks 2 and 7 at the PEAK Laboratory at the URMC (see Section 6.7).

5.4 An optional fasting (8-hour) blood draw will be done at the URMC to estimate cytokines (CRP, IL-6, & TNF-α) during study weeks 2 and 7 (see Section 6.8).

5.5 Treatment Arms:

5.5.1 Subjects assigned to Arm 1 will receive two massage treatments approximately two weeks apart.

5.5.2 Subjects assigned to Arm 2 will receive two Reiki treatments approximately two weeks apart.

5.5.3 Subjects assigned to Arm 3 will receive four Reiki treatments approximately 1 week apart.

5.5.4 Scheduling arrangements will be made for the treatments prior to the initiation of the intervention.

5.5.6 Subjects will not be charged for the Reiki or massage treatments.

ELIGIBILITY:
Inclusion Criteria:

* Be a breast cancer patient receiving an aromatase inhibitor (AI) and not be scheduled to have a change in treatment during the next 10 weeks or have prostate cancer and be on a stable dose of ADT for at least 8 weeks and not be scheduled to have a change in treatment during the next 10 weeks.
* Be at least two months out from the conclusion of any prior surgery, chemotherapy, radium 223 therapy, abiraterone, enzalutamide, Sipuleucel-T, or radiation therapy.
* Have a response of 4 or greater on a question assessing fatigue at its worst during the past week that is assessed on an 11-point scale anchored by "0" = no fatigue and "10" = worst possible fatigue.
* Be able to read English (since the assessment materials will be in a printed format).

Exclusion Criteria:

* Be scheduled to receive surgery, chemotherapy, radium 223 therapy, abiraterone, enzalutamide, Sipuleucel-T, or radiation therapy during the next 10 weeks.
* Be taking erythropoietin or darbepoetin for anemia.
* Have received Therapeutic Touch, Reiki, Polarity Therapy, or professional massage therapy during the prior four weeks.
* Have a bleeding disorder, blood clot, previous neck/back injury, or other medical condition that would, in the estimation of their physician (or their designee), preclude having massage therapy.

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 87 (Actual)
Dates: Start 2016-06-20 (Actual); Primary Completion 2019-04 (Actual); Study Completion 2019-05 (Actual)

PRIMARY OUTCOMES:
The revised Brief Fatigue Inventory (BFI) | The primary outcome measure for this study is fatigue assessed on Friday during study week 6 by the BFI.
  The revised Brief Fatigue Inventory (BFI) is a 9-item, patient-report instrument with established reliability and validity.

CONTACTS AND LOCATIONS:
Overall Officials: Luke Peppone, Ph.D., Principal Investigator — University of Rochester
Locations (1):
- University of Rochester Wilmot Cancer Institute, Rochester, New York, United States

IPD SHARING:
Plan to Share IPD: No